CLINICAL TRIAL: NCT01642654
Title: Nitrite Levels and Vascular Function in Elderly Women Submitted to Water Exercise: a Randomised Controlled Trial
Brief Title: Water Exercise and Vascular Function in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Yula Pires da Silveira Fontenele de Meneses, Msc, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: yula01
Record Dates: First submitted 2012-07-10; First posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-03

CONDITIONS: Elderly Women
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator)
  Interventions: Other: Educational lectures
- Treatment (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The WG was submitted to a 16-week WEP, with combined aerobic and resistance exercises in three weekly sessions. Water temperature was approximately 30º C with an average ambient temperature of 34° C. The pool had water levels ranging between 1,20 and 1,40 meters deep.
  Arms: Treatment
Other: Educational lectures — Educational lectures
  Arms: Control

SUMMARY:
Objectives:

The purpose of this research was to assess modifications caused by a concurrent water exercise program on plasma nitrite (NO3), cerebral vascular resistance and cholesterol in the elderly and analyze the correlations between these variables after intervention.

Methods The sample was composed of 40 women mean age 69,21 ±5,27 years old, divided into an intervention (WG) and control group (CG). It was to measure nitrite concentration (NO3) by the Griess reaction; internal cerebral arteries were assessed by Doppler ultrasound to determine the resistivity index and Cholesterol was determined using the colorimetric enzymatic method and test kit. Intervention with water exercise program consisted of three weekly sessions for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* older than 60 and lass than 80 years age;
* the elderly should be independent in their ADLs;
* be considered able for medical evaluation to participate in the intervention and testing protocols;
* still not be participating in regular systematized physical activity for at least six months.

Exclusion Criteria:

* subjects with any form of transmittable or uncontrolled disease or insulin-dependent hypertensive;
* unable to perform functional autonomy tests;
* women undergo hormonal replacement therapy

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Determining modifications caused by this program on plasma nitrite concentration (NO3). | 16 weeks
  For NO analysis, serum was separated from the erythrocyte mass. The material was centrifuged in a SIGMA 4k15 centrifuge at 3500 rpm and 18° for 10 minutes (LANEX laboratory- UFPI); the serum was then pipetted and frozen at 80° for evaluation after retesting (16 weeks). NO production was determined based on NO3 in the supernatant of cultured cells, an indirect measurement of NO synthesis.

SECONDARY OUTCOMES:
Cerebral artery assessment | 16 weeks
  Carotid and vertebral arteries were assessed by Doppler ultrasound, with GE Logiq 5 equipment and multi-frequency linear transducer (Milwaukee - UEA). Parameters used were evaluation of peak systolic velocity and end-diastolic velocity of the common carotid and left and right internal carotids, with the angle of insonation corrected to 60°. The resistivity index of arteries was calculated, resulting from the mathematical formula in centimeters per second (cm/s): Resistivity index = Peak systolic velocity - End-diastolic velocity / Peak systolic velocity.

CONTACTS AND LOCATIONS:
Overall Officials: Arméle Dornelas, Study Chair — Universidade Federal de Pernambuco
Locations (1):
- Universidade Estadual do Piauí, Teresina, Piauí, Brazil

REFERENCES:
- [Result] Cress ME, Buchner DM, Prohaska T, Rimmer J, Brown M, Macera C, Dipietro L, Chodzko-Zajko W. Best practices for physical activity programs and behavior counseling in older adult populations. J Aging Phys Act. 2005 Jan;13(1):61-74. doi: 10.1123/japa.13.1.61. PMID 15677836